CLINICAL TRIAL: NCT01166035
Title: Phase 1/2 Study of Lenalidomide and Cetuximab in Patients With Advanced Solid Tumors
Brief Title: Lenalidomide and Cetuximab in Patients With Advanced Solid Tumors
Acronym: TEXO
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Celgene Corporation (Industry); Innsbruck - Tyrolean Working Group of Experimental Oncology (TEXO) (Unknown)
Responsible Party: Medical University of Innsbruck, Department of Internal Medicine I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEXO0309
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-05

CONDITIONS: Solid Tumors
Keywords: Solid tumors; Lenalidomide; Cetuximab; Colorectal Cancer; Non-Small Cell Lung Cancer; Head and Neck Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms | interventions — Lenalidomide; Cetuximab

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide will be supplied as 5 mg, 10 mg, 15 mg, 20 mg and 25 mg capsules for oral administration.
  Prior to Cycle 1, there will be a 21 day lead in treatment period with lenalidomide monotherapy (Days -21 to -1). Combination treatment will start at Day 1. Subjects will be enrolled in cohorts of three to receive a single, oral dose of lenalidomide administered on Days 1-28. For each cohort of subjects, the decision of whether or not to dose-escalate will be made after subjects have received the first treatment cycle of study drug. Treatment will continue until the occurrence of any of the following events.
  * Disease progression
  * Adverse event(s) that, in the judgment of the Investigator, may cause severe or permanent harm or which rule out continuation of the treatment regimen.
  * Major violation of the study protocol.
  * Withdrawal of consent
  * Lost to follow up
  * Death
  * Suspected pregnancy
Drug: Cetuximab — Combination treatment will start at Day 1. Subjects meeting will be enrolled in cohorts of three to receive infusions of cetuximab (400 mg/m2 first infusion only, then 250 mg/m2 subsequently) administered on Days 1, 8, 15, and 22 of each 28-day cycle. Cetuximab will be supplied as Erbitux® 22 mg/ml Vial à 50 ml, Erbitux 5 mg/ml Vial à 10 ml and Erbitux 5 mg/ml Vial à 50 ml for intravenous administration.
  Treatment will continue until the occurrence of any of the following events.
  * Disease progression
  * Adverse event(s) that, in the judgment of the Investigator, may cause severe or permanent harm or which rule out continuation of the treatment regimen.
  * Major violation of the study protocol.
  * Withdrawal of consent
  * Lost to follow up
  * Death
  * Suspected pregnancy

SUMMARY:
This is a Phase 1/2, open-label, monocentric, dose-escalation study of lenalidomide in combination with cetuximab in subjects with solid tumors. The primary objective is to establish the maximum tolerated dose (MTD) of lenalidomide in combination with cetuximab in patients with solid tumors including colorectal cancer (CRC), squamous cell carcinoma of the head and neck (SCCHN) and non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Background: For metastatic cancer such as head and neck, lung and colorectal cancer, standard therapy comprises chemotherapy regimen partially in combination with monoclonal antibodies blocking the vascular endothelial growth factor (VEGF) or the epidermal growth factor receptor (EGFR). When disease progression occurs during or after these treatment options have been applied, no established therapy is available and the clinical development of new strategies is warranted. Lenalidomide (Revlimid®) is a thalidomide derivative and belongs to the so-called ImiDs, a class of immunostimulatory molecules. IMiDs have profound effects on the immune system. Obviously, IMiDs are able to function as co-stimulatory molecule for mature T cells. In addition, IMiDs are able to mitigate the negative effects of CTLA-4 signalling. On the molecular level, IMiDs induce phosphorylation of CD28, underlining the concept that they act as costimulatory signals during T cell activation. Furthermore, the induction of specific CTL responses by dendritic cells (DC) is enhanced and the activity of suppressive regulatory T cells (Treg) inhibited.

In addition to their effects on cells of the adaptive immune system, IMiDs also target the innate immune response. Natural killer cells (NK) as well as natural killer T-cells (NKT) are activated by Immunomodulatory Drugs (IMiDs), and the effects of IMiDs on NK and NKT cells might further contribute to the immune-activating properties of ImiDs.

Therefore the rationale of the combination of lenalidomide with a therapeutic IgG1 antibody such as cetuximab (Erbitux®) is based on the fact that several reports suggest a role of antibody-dependent cellular cytotoxicity (ADCC) as a mode of action of cetuximab.

However, the exact definition of these anti-cancer mechanisms of lenalidomide alone and in combination with cetuximab in vivo require further investigation in early clinical trials.

The goal of this phase I/II trial is to define the toxicity of the combination of lenalidomide and cetuximab and to study potential effects on the tumor and the immune system.

Subjects meeting all inclusion criteria will be enrolled in cohorts of three patients to receive a single, oral dose of lenalidomide administered on Days 1-28 and intravenous (IV) infusions of cetuximab (400 mg/m2 first infusion only, then 250 mg/m2 subsequently) administered on Days 1, 8, 15, and 22 of each 28-day cycle.

Prior to combination therapy, there will be a 21 day lead in treatment period with lenalidomide monotherapy (Days -21 to -1). Combination treatment will start at Day 1. Tumor biopsies will be taken before monotherapy lenalidomide treatment (between d-25 and -22) and between Day -3 and -1 (before starting cetuximab). A third tumor biopsy will be taken between Cycle 1 Day 21 and 28 after starting combination therapy. Cycles will be repeated every 28 days. All subjects will continue on study drug until disease progression, unacceptable toxicity or treatment discontinuation for any other reason. The MTD of lenalidomide will be defined as the highest dose level at which no more than 1 out of 6 subjects experience a dose-limiting toxicity (DLT) during the first cycle of administration in combination with cetuximab. Safety measurements and analysis will be performed at each visit.

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics:

1. Patients signed informed consent.
2. Histologically or cytologically confirmed SCCHN, NSCLC, or metastatic colorectal adenocarcinoma.
3. At least one unidimensionally measurable lesion.
4. 18 - 80 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of <= 1.
6. Female subjects of childbearing potential must:

   * Understand that the study medication could have an expected teratogenic risk
   * Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea. An alternative would be an absolute and continued sexual abstinence.

   The following are effective methods of contraception*
   * Implant
   * Levonorgestrel-releasing intrauterine system (IUS)**
   * Medroxyprogesterone acetate depot
   * Tubal sterilisation
   * Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses Ovulation inhibitory progesterone-only pills (i.e., desogestrel)

     * Combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of VTE continues for 4 to 6 weeks after stopping combined oral contraception.
     * Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days before the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
     * Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start
   * of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence
7. Male subjects must

   * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
   * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
8. All subjects must

   * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
   * Agree not to share study medication with another person and to return all unused study drug to the investigator

Exclusion Criteria:

Prior Treatment:

1. Use of chemotherapy, hormonal therapy, immunotherapy, or any other anticancer or experimental therapy within 28 days prior to study medication.
2. Active participation in another clinical trial.
3. Radiotherapy within 28 days prior to study medication.
4. Surgery within 28 days prior to study medication (minimally invasive procedures for the purpose of diagnosis or staging of the disease are permitted).
5. Prior therapy with pomalidomide (CC-4047), lenalidomide, or thalidomide.

   Laboratory:
6. Absolute neutrophil count (ANC) < 1.5 x 109/L.
7. Platelet count < 100 x 109/L.
8. Creatinine Clearance < 50 mL/min.
9. Bilirubin > 1.5 x Upper Limit Normal (ULN) (> 2.0 x ULN in the presence of Gilbert's Syndrome).
10. Serum aspartate transaminase (AST)/SGOT > 3.0 x ULN (> 5 x ULN in the presence of liver metastases).

    Other Disease State:
11. Untreated, symptomatic brain metastases (brain imaging not required).
12. Venous thromboembolism within 6 months.
13. Current congestive heart failure (New York Heart Association class II-IV).
14. Uncontrolled hypertension
15. Prior malignancies within 5 years, with the exception of treated basal cell/squamous cell carcinoma of the skin or "in-situ" carcinoma of the cervix or breast.

    General:
16. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study or confound the ability to interpret data from the study.
17. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
18. Pregnant or lactating females.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | on the end of every treatment cycle (28 day-cycles).
  Determination of the maximum tolerated dose (MTD) of lenalidomide administered in combination with cetuximab. For each cohort of subjects (3 patients), the decision of whether or not to dose-escalate will be made after subjects have received the first treatment cycle of study drug. Once 2 subjects have experienced DLT, enrollment at that dose will end and that dose will be declared to have exceeded the MTD.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Zwierzina, Prof. Dr., Principal Investigator — Medical University of Innsbruck, Deparmtment of Internal Medicince I
Locations (1):
- Medical University of Innsbruck, Department for Internal Medicine I, Innsbruck, Tyrol, Austria

REFERENCES:
- [Derived] Gamerith G, Auer T, Amann A, Putzer D, Schenk B, Kircher B, Hilbe W, Zwierzina H, Loeffler-Ragg J. Increase in antibody-dependent cellular cytotoxicity (ADCC) in a patient with advanced colorectal carcinoma carrying a KRAS mutation under lenalidomide therapy. Cancer Biol Ther. 2014 Mar 1;15(3):266-70. doi: 10.4161/cbt.27327. Epub 2013 Dec 18. PMID 24351336